CLINICAL TRIAL: NCT02098382
Title: Prospective Collection of Data About the Use of the Dilapan-S Osmotic Dilator in Pre-induction of Labor in Women With/Without Caesarean Section in Their History
Brief Title: Dilapan-S Osmotic Dilator in Pre-induction of Labor
Status: Completed | Type: Observational
Sponsor: Medicem International CR s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: DIS2013-002
Record Dates: First submitted 2014-03-10; First posted 2014-03-28 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2014-03

CONDITIONS: Uterine Cervical Incompetence
Keywords: Cervical ripening
MeSH Terms: conditions — Uterine Cervical Incompetence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dilapan-S: 125 Patients with / without caesarean section in their medical history
  Interventions: Device: Dilapan-S

INTERVENTIONS:
Device: Dilapan-S — Dilapan-S synthetic osmotic dilator for cervical ripening prior to labor induction
  Other Names: synthetic osmotic dilator

SUMMARY:
Non-interventional prospective data collection designed to evaluate clinical outcome on the efficacy of the use of Dilapan-S in the indication of labor pre-induction in women with/without a history of Caesarean section. The evaluation will be based on prospective data collection in at least four obstetrics centers in the Czech Republic.

DETAILED DESCRIPTION:
Nowadays there is a rising need for non-pharmacological cervical ripening methods as the use of prostaglandins is frequently limited by various contraindications. Dilapan-S is a hygroscopic uterine neck dilator. Its mode of action consists in the hydrophilic properties of the device absorbing fluids from surrounding tissue structures, thus expanding the volume of Dilapan-S sticks which subsequently exert radial pressure on the surrounding structures (uterine neck) to dilate progressively. Endocervical pressure on the uterine neck results not only in its mechanical dilatation but pressure on endocervical structures also stimulates the production of endogenous prostaglandins, which promote cervical ripening through its collagenolytic action. Although Dilapan-S is widely used in labor pre-induction, published study data comparing its clinical efficacy and safety in females with/without caesarean section in medical history are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Pregnancy more than 36 weeks
* Vertex presentation of the fetus
* Cervix Score less than 4 points

Exclusion Criteria:

* Contraindication to vaginal delivery
* Pathological fetal station
* States after uterine body surgery - except for Caesarean section
* Clinical signs of uterine, vaginal or vulvar infection
* Fetus hypoxia (KTG recording evaluated as pathological prior to pre-induction initiation)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients indicated in the centres involved in data collection for pre-induction of labor with Dilapan-S who meet all inclusion and exclusion criteria.
  In the above period, the Investigator will include consecutive patients in such a manner that the numbers of those with and without a history of Caesarean section be balanced.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cervix (Bishop) score | Before pre-induction of labor performance and up to 24 h after pre-induction of labor
  To evaluate, based on the value obtained in the Cervix Score, the efficacy of use of the Dilapan-S device in the indication labor pre-induction, and to compare outcomes in patients with/without a history of Caesarean section.

SECONDARY OUTCOMES:
Total duration of pre-induction | From Dilapan-S rods insertion up to 24 hours
  To compare these outcomes in patients with and without a history of Caesarean section.
Number of dilators inserted | At the moment of Dilapan-S insertion up to 24 hours until their removal
  Expected the insertion from 2 to 5 Dilapan-S rods. To compare these results in patients with/without Cesarean section in their medical history.
Uterine contractions | From Dilapan-S rods insertion up to 24 h during pre-induction of labor phase
  To compare these results in patients with/without Caesearean section in their medical history. Uterine hypertonus is diagnosed, when the number of uterine contractions is higher than 5 within 10 minutes (during pre-induction).
The course of delivery (vaginally or Caesarean section) | From active phase of labor up to 1 day after delivery
  To compare the rate of vaginal delivery/Caesarean sections in patients with/without Caesarean section in their medical history.
Apgar score | At 1st, 5th and 10th minute after delivery
  To compare these results in patients with/without Caesarean section in their medical history.
pH of the fetus | Up to 10 minutes after delivery
  To compare the results in patients with/without caesarean section in their medical history. The rate of ceses with pH below 7,1.
Infection complications of mother / fetus | Up to 5 days from the birth
  Clinical signs of infection are defined as follows:
  1. CRP levels > 8 mg/l
  2. Leukocyte count > 18 x 109/l
  3. Body temperature > 37.5°C

OTHER OUTCOMES:
Course of removal of Dilapan-S rods after pre-induction | At the moment of removal of Dilapan-S rods after labor pre-induction phase up to 1 day after delivery
  The evaluation of the course of removal of Dilapan-S after termination of preinduction by physician as very easy, easy, standard, with some complications or very complicated.
Occurance of complication of rupture of fetal sac due to the use of Dilapan-S or other complications related to the use of Dilapan-S | From Dilapan-S rods insertion up to 24 h of duration of labor pre-induction phase
Patients´evaluation of pre-induction of labor with Dilapan-S | From Dilapan-S insertion up to 24 h of duration of labor pre-induction phase
  Subjective satisfaction Pain experienced during Dilapan-S insertion and pre-induction phase Quality of relax and sleep Frequency and intensity of uterine contractions during pre-induction

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Simetka, AssProf,PhD, Principal Investigator — Clinic of gynecology and obstetrics, University hospital of Ostrava, Czech Republic; Lukas Hruban, M.D., Principal Investigator — Clinic of gynecology and obstetrics, University hospital of Brno, Czech Republic; Igor Michalec, M.D., Principal Investigator — Clinic of gynecology and obstetrics, University hospital of Ostrava, Czech Republic; Radovan Vlk, M.D., Principal Investigator — Clinic of gynecology and obstetrics, University hospital of II. Medicine college of Charles University in Prague, Czech Republic
Locations (1):
- Clinic of Gynecology&Obstetrics, University hospital in Brno and Masaryk University Medical School, Brno, Czechia

REFERENCES:
- [Background] Serhal P, Ranieri DM, Khadum I, Wakim RA. Cervical dilatation with hygroscopic rods prior to ovarian stimulation facilitates embryo transfer. Hum Reprod. 2003 Dec;18(12):2618-20. doi: 10.1093/humrep/deg477. PMID 14645181
- [Background] Chen FC, Bergann A, Krosse J, Merholz A, David M. Isosorbide mononitrate vaginal gel versus misoprostol vaginal gel versus Dilapan-S for cervical ripening before first trimester curettage. Eur J Obstet Gynecol Reprod Biol. 2008 Jun;138(2):176-9. doi: 10.1016/j.ejogrb.2007.09.009. Epub 2007 Nov 5. PMID 17980952
- [Background] Allen RH, Goldberg AB; Board of Society of Family Planning. Cervical dilation before first-trimester surgical abortion (<14 weeks' gestation). SFP Guideline 20071. Contraception. 2007 Aug;76(2):139-56. doi: 10.1016/j.contraception.2007.05.001. Epub 2007 Jul 10. PMID 17656184
- [Background] Samuel MI, Parsons JH. Hygroscopic dilator (Dilapan-S) and misoprostol combination for the early first-trimester termination of pregnancy: a pilot study. J Fam Plann Reprod Health Care. 2009 Jan;35(1):45-7. doi: 10.1783/147118909787072234. PMID 19126319
- [Background] Wilson LC, Meyn LA, Creinin MD. Cervical preparation for surgical abortion between 12 and 18 weeks of gestation using vaginal misoprostol and Dilapan-S. Contraception. 2011 Jun;83(6):511-6. doi: 10.1016/j.contraception.2010.10.004. Epub 2010 Dec 3. PMID 21570547
- [Background] Chambers DG, Willcourt RJ, Laver AR, Baird JK, Herbert WY. Comparison of Dilapan-S and laminaria for cervical priming before surgical pregnancy termination at 17-22 weeks' gestation. Int J Womens Health. 2011;3:347-52. doi: 10.2147/IJWH.S25551. Epub 2011 Oct 20. PMID 22114527
- [Background] Lyus R, Lohr PA, Taylor J, Morroni C. Outcomes with same-day cervical preparation with Dilapan-S osmotic dilators and vaginal misoprostol before dilatation and evacuation at 18 to 21+6 weeks' gestation. Contraception. 2013 Jan;87(1):71-5. doi: 10.1016/j.contraception.2012.07.006. Epub 2012 Aug 13. PMID 22898362
- [Background] Fox MC, Krajewski CM. Cervical preparation for second-trimester surgical abortion prior to 20 weeks' gestation: SFP Guideline #2013-4. Contraception. 2014 Feb;89(2):75-84. doi: 10.1016/j.contraception.2013.11.001. Epub 2013 Nov 11. PMID 24331860
- [Background] Bartz D, Maurer R, Allen RH, Fortin J, Kuang B, Goldberg AB. Buccal misoprostol compared with synthetic osmotic cervical dilator before surgical abortion: a randomized controlled trial. Obstet Gynecol. 2013 Jul;122(1):57-63. doi: 10.1097/AOG.0b013e3182983889. PMID 23743471
- [Background] Borgatta L, Roncari D, Sonalkar S, Mark A, Hou MY, Finneseth M, Vragovic O. Mifepristone vs. osmotic dilator insertion for cervical preparation prior to surgical abortion at 14-16 weeks: a randomized trial. Contraception. 2012 Nov;86(5):567-71. doi: 10.1016/j.contraception.2012.05.002. Epub 2012 Jun 6. PMID 22682721
- [Background] Borgatta L, Lopatinsky I, Shaw FM. Overcoming unsatisfactory colposcopy. Use of osmotic dilators. J Reprod Med. 1997 May;42(5):271-5. PMID 9172116
- [Background] Newmann SJ, Sokoloff A, Tharyil M, Illangasekare T, Steinauer JE, Drey EA. Same-day synthetic osmotic dilators compared with overnight laminaria before abortion at 14-18 weeks of gestation: a randomized controlled trial. Obstet Gynecol. 2014 Feb;123(2 Pt 1):271-278. doi: 10.1097/AOG.0000000000000080. PMID 24402587
- [Result] Roztocil A, Pilka L, Jelinek J, Koudelka M, Miklica J. A comparison of three preinduction cervical priming methods: prostaglandin E2 gel, Dilapan S rods and Estradiol gel. Ceska Gynekol. 1998 Feb;63(1):3-9. PMID 9650373